CLINICAL TRIAL: NCT03791216
Title: Characterization of Lipoprotein Composition and Function in Pediatric Psoriasis Before and After Treatment
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Psoriasis Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital of Philadelphia (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Other Study IDs: 2019-2361
Record Dates: First submitted 2018-12-05; First posted 2019-01-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for lipids testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Psoriasis patients to be treated only topically
  Interventions: Other: Fasting blood draw for lipid assessments
- Psoriasis patients with moderate-to-severe psoriasis who begin
  Interventions: Other: Fasting blood draw for lipid assessments
- Age-, sex- and BMI percentile-matched controls
  Interventions: Other: Fasting blood draw for lipid assessments
- Patients being treated with isotretinoin for acne
  Interventions: Other: Fasting blood draw for lipid assessments

INTERVENTIONS:
Other: Fasting blood draw for lipid assessments — Fasting blood draw for lipid assessments

SUMMARY:
This study will assess differences in inflammatory proteins, lipoprotein composition, cholesterol efflux and HDL-proteome in moderate-to-severe pediatric psoriasis who at baseline begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6-17 years of all races/ethnicities with plaque and/or extensive guttate psoriasis for at least 6 months and on topical or systemic therapy
* Patients in the systemic group can be starting a medication for the first time OR transitioning from another systemic if unresponsive and on that previous treatment for ≤ 3 months.
* Patients may concurrently have psoriatic arthritis if initiation of a systemic medication is warranted by skin severity.
* Children ages 6-17 years of all races/ethnicities with acne being treated with isotretinoin
* Children ages 6-17 years of all races/ethnicities without plaque or guttate psoriasis and history of severe acne or treatment with isotretinoin as controls.

Exclusion Criteria:

* Patients less than 6 years of age or 18 years and older
* Patients with congenital heart disease, prior cardiac catheterizations/surgeries, or on cardiac medications in the past two years other than for hypertension (eg, calcium channel-blockers, beta-blockers and vasotropic medications).
* Patients who have other systemic inflammatory diseases (including atopic dermatitis, severe acne, inflammatory bowel disease, juvenile idiopathic arthritis, connective tissue diseases and/or other autoimmune diseases).
* Patients who have active infection or malignancy or have suffered from infection requiring oral or parenteral antibiotic in past 2 weeks.
* Patients and parents/caregivers unable to give written informed consent.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators plan to recruit approximately 120 subjects total. Subjects will be divided into 4 groups: i) patients to be treated only topically (n=30); ii) patients with moderate-to-severe psoriasis who begin systemic treatment (n=30; ~15 DMARDs and 15 biologics); iii) age-, sex- and BMI percentile-matched controls (n=30); iv) patients being treated with isotretinoin for acne (n=30).
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Lipoprotein composition differences-glucose | one year
  To assess differences in the blood concentration levels at baseline for glucose in moderate-to-severe pediatric psoriasis at baseline who begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.
Lipoprotein composition differences-insulin | one year
  To assess differences in the blood concentration levels at baseline for insulin in moderate-to-severe pediatric psoriasis at baseline who begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.
Lipoprotein composition differences-c-reactive protein | one year
  To assess differences in the blood concentration levels at baseline for c-reactive protein in moderate-to-severe pediatric psoriasis at baseline who begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.
Lipoprotein composition differences-lipid concentration | one year
  To assess differences in the blood concentration levels at baseline for lipid concentration in moderate-to-severe pediatric psoriasis at baseline who begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.
Lipoprotein composition differences-chemistry panel | one year
  To assess differences in the blood concentration levels at baseline for chemistry panel in moderate-to-severe pediatric psoriasis at baseline who begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.
Lipoprotein composition differences-apolipoprotein | one year
  To assess differences in the blood concentration levels at baseline for apolipoprotein in moderate-to-severe pediatric psoriasis at baseline who begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.
Lipoprotein composition differences-NMR | one year
  To assess differences in the blood concentration levels at baseline for NMR derived lipoprotein particle concentrations in moderate-to-severe pediatric psoriasis at baseline who begin systemically administered therapy vs: a) healthy controls; and b) patients with milder psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No